CLINICAL TRIAL: NCT02639468
Title: Electric Impedance Tomography
Acronym: SVEIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol not fully appropriate technical issues with EIT device
Sponsor: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SVEIT
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Stroke Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tomographie par impédance électrique (Experimental): Tomographie par impédance électrique
  Interventions: Device: Stroke Volume estimation using electrical impedance tomography

INTERVENTIONS:
Device: Stroke Volume estimation using electrical impedance tomography

SUMMARY:
Evaluation of electrical impedance tomography to non-invasively monitor stroke volume when compared to reference measurements performed via right heart thermodilution

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery which requires placement of pulmonary catheter
* Patients with right heart catheterization for diagnostic or therapeutic reasons

Exclusion Criteria:

* Patient unable to understand the study
* Patient unable to provide written consent or refusing his/her participation
* Patient suffering from a severe valvular insufficiency
* Patient allergic to ECG electrodes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Correlation of stroke volume values measured via pulmonary catheter compared to EIT-derived stroke volume estimates. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No